CLINICAL TRIAL: NCT01395628
Title: Xenotransplantation of Primary Leukemia Samples Into Zebrafish
Brief Title: Cell Samples From Patients With Leukemia
Status: Completed | Type: Observational
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: AAML11B13; COG-AAML11B13 (Other: Children's Oncology Group); AAML11B13 (Other: Children's Oncology Group); NCI-2011-02863 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2011-07-14; First posted 2011-07-15 (Estimated); Last update posted 2016-05-19 (Estimated); Status verified 2016-05

CONDITIONS: Leukemia
Keywords: chronic phase chronic myelogenous leukemia; childhood acute promyelocytic leukemia (M3); childhood acute myeloid leukemia/other myeloid malignancies; adult acute myeloid leukemia with t(8;21)(q22;q22); adult acute myeloid leukemia with del(5q); adult acute promyelocytic leukemia (M3)
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid, Chronic-Phase; Leukemia, Promyelocytic, Acute | interventions — Flow Cytometry; Microscopy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — cell samples
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: in vitro sensitivity-directed chemotherapy
Other: cell proliferation assay
Other: fluorescence activated cell sorting
Other: laboratory biomarker analysis
Other: microscopy

SUMMARY:
RATIONALE: Studying samples of blood and tissue from patients with cancer in the laboratory may help doctors learn more about cancer and the development of drug resistance in patients. It may also help doctors find better ways to treat cancer.

PURPOSE: This research trial is studying samples from patients with leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* Demonstrate the capability of primary human leukemia samples to survive and proliferate in the zebrafish embryo.
* Confirm the anti-proliferative or toxic effects of known chemotherapeutics on the transplanted cells in vivo.
* Evaluate the effect of novel anticancer drugs and/or their combinations on individual samples.

OUTLINE: This is a multicenter study.

Cryopreserved specimens are injected into the yolk sac of zebrafish embryos under anesthesia. After 1 hour of recovery at 28° C, embryos are maintained at 38° C and screened for fluorescence at the injection site. Within 48 hours post-injection, some embryos are treated with various chemotherapeutic drugs or dimethyl sulfoxide and incubated in protease solution. Proliferation of leukemia cells are monitored by live-cell microscopy. Cells with or without drug treatment are then extracted at 24 and 72 hours post-injection. Leukemia cells are counted and tested with imatinib mesylate, all-trans retinoic acid (tretinoin), cytosine arabinose, and known bioactive chemical compounds from promising drug families, such as tyrosine kinase inhibitors, antiapoptotic agents, channel modulators, and prostaglandin agonists.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Samples of blood and tissue cells from patients diagnosed with myeloid disease including the following subtypes:

  * Chronic phase chronic myeloid leukemia (CML), to complement initial studies in the K562 CML cell line
  * Acute promyelocytic leukemia (APL), to complement initial studies in the NB4 APL cell line
  * Acute myeloid leukemia (AML) expressing the t(8;21)(q22;q22) translocation, which occurs in approximately 12% of pediatric AML and is associated with good prognosis
  * AML expressing 5q- or monosomy 7, associated with a poor prognosis
  * AML expressing the fms-like tyrosine kinase 3 internal tandem duplication (FLT3-ITD), associated with a poor prognosis

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* Not specified

Max Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients diagnosed with myeloid disease.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2011-07; Primary Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Primary human leukemia samples capable to survive and proliferate in the zebrafish embryo
In vivo confirmation of anti-proliferative or toxic effects of known chemotherapeutic agents on the transplanted cells
Effects of novel anticancer drugs and/or their combinations on individual samples

CONTACTS AND LOCATIONS:
Overall Officials: Jason N. Berman, MD, Principal Investigator — IWK Health Centre